CLINICAL TRIAL: NCT04965623
Title: ExplorATory Study oF the EdWards Transcatheter Atrial Shunt System (AlT FloW Germany)
Acronym: AlT-FloW
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was not initiated due to Covid. Then, Edwards Lifesciences elected to withdraw this study due to the initiation of the ALT-FLOW II randomized trial in Germany.
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-14
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Edwards Transcatheter Atrial Shunt System (Experimental): Edwards Transcatheter Atrial Shunt System
  Interventions: Device: Atrial Shunt

INTERVENTIONS:
Device: Atrial Shunt — Transcatheter treatment of symptomatic left heart failure patients

SUMMARY:
The Exploratory Study of the Edwards Transcatheter Atrial Shunt System is a multi-center, prospective, exploratory study to evaluate initial clinical safety, device functionality, and effectiveness of the Edwards Transcatheter Atrial Shunt System.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Ethics Committee (EC) approved study consent form prior to study related procedures
2. ≥ 18 years old
3. Chronic symptomatic Heart Failure (HF) documented by the following:

   1. NYHA class III or ambulatory NYHA class IV within last 12 months AND
   2. ≥ 1 HF hospital admission (with HF as the primary, or secondary diagnosis); or treatment with intravenous (IV) or intensification of oral diuresis for HF in a healthcare facility (emergency department/acute care facility) within the 12 months prior to study entry; OR an NT-pro BNP value > 150 pg./ml in normal sinus rhythm, > 450 pg./ml in atrial fibrillation, or a BNP value > 50 pg./ml in normal sinus rhythm, > 150 pg./ml in atrial fibrillation within the past 6 months.
4. In the judgment of the investigator, subject is on stable Guideline Directed Medical Therapy (GDMT) for heart failure and management of potential comorbidities according to current ACCF/AHA/ESC Guidelines and that is expected to be maintained without change for 3 months
5. Elevated LA (or PCWP) pressure of > 15 mmHg at rest or > 25 mmHg during supine ergometer exercise stress test, as measured at end-expiration; AND the LA (or PCWP) exceeds right atrial pressure (RAP) by > 5 mmHg at rest or > 10 mmHg during supine ergometer exercise stress test as measured at end-expiration
6. Willing to attend study follow-up assessments for up to 5 years

Exclusion Criteria:

1. Severe heart failure defined as one or more of the below:

   1. ACC/AHA/ESC Stage D heart failure, non-ambulatory NYHA Class IV HF
   2. If BMI < 30, Cardiac index < 2.0 L/min/m2
   3. If BMI ≥ 30, cardiac index < 1.8 L/min/m2
   4. Inotropic infusion (continuous or intermittent) within the past 6 months
   5. Patient is on the cardiac transplant waiting list
   6. LVEF < 20%
2. Presence of significant valve disease defined by the site cardiologist as:

   1. Mitral valve regurgitation defined as grade > 3+ MR or > moderate MS
   2. Tricuspid valve regurgitation defined as grade > 2+ TR
   3. Aortic valve disease defined as > 2+ AR or > moderate AS
3. MI and/or any therapeutic invasive cardiac procedure within past 3 months; or current indication for coronary revascularization
4. Valve replacement or surgical annuloplasty within the past 12 months
5. Stroke or transient ischemic attack (TIA) within the past 6 months
6. Hemodynamic instability within 30 days of scheduled implant procedure
7. Patient requiring surgery under general anesthesia for any reason within 30 days of scheduled implant procedure
8. Clinically diagnosed hypertrophic obstructive cardiomyopathy, constrictive pericarditis or other infiltrative cardiomyopathy (eg, hemochromatosis, sarcoidosis) at the time of screening per central screening committee
9. Has renal insufficiency as determined by creatinine (S-Cr) level > 2.5 mg/dL or estimated-GFR < 25ml/min/1.73 m2 by CKD-Epi equation; or currently requiring dialysis
10. Significant hepatic impairment defined as 3× upper limit of normal of transaminases, total bilirubin, or alkaline phosphatase
11. Right ventricular dysfunction, defined by the site cardiologist as:

    1. More than mild RV dysfunction as estimated by TTE; OR
    2. TAPSE <1.4 cm; OR
    3. RV size ≥ LV size as estimated by TTE; OR
    4. Echocardiographic or clinical evidence of congestive hepatopathy;
12. Evidence of pulmonary hypertension with PVR >4 Wood units
13. Performance of the 6 minute walk test with a distance <50m OR >600m
14. Subject is contraindicated to receive either dual antiplatelet therapy or warfarin (analogue); or has a documented coagulopathy
15. Known hypersensitivity to anticoagulation therapy or contrast agent, which cannot be adequately medicated
16. Known hypersensitivity to Nickel and/or Tantalum
17. In the judgment of the investigator, life expectancy <12 months for noncardiovascular reasons
18. In the opinion of the investigator and Central Screening Committee, the subject is not an appropriate candidate for the study
19. Anatomy or implantable device that is not compatible with or could potentially interfere with the Edwards Transcatheter Atrial Shunt System as determined by the Investigator and Central Screening Committee
20. Active endocarditis or infection within 3 months of scheduled implant procedure
21. Currently participating (e.g., undergoing trial specific exams/treatment/procedures) in an investigational drug or device study. Note: trials requiring extended follow-up for products that were investigational but have since become commercially available are not considered investigational trials.
22. Patient is a current intravenous drug user
23. Positive serum pregnancy test in female subjects of child-bearing potential or nursing mothers or planning on becoming pregnant during the duration of the trial
24. Patient is under guardianship
25. Known pre-existing shunting, determined to be clinically significant by the investigator and Central Screening Committee
26. Patients with a CRT lead in the coronary sinus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Rate of Safety Events (MACCREE, Re-Intervention) | 30 Days
  Composite of major adverse cardiac, cerebrovascular, renal events (MACCRE) and re-intervention for study device related complications at 30 days.

SECONDARY OUTCOMES:
Rate of Device Success | Day 0
  Device is deployed as intended and the delivery system is successfully removed as intended at the time of the patient's exit from the implant procedure room.
Rate of Procedural Success | 10 Days post-op
  Device success with evidence of shunt patency and hospital discharge without the need for additional surgical or percutaneous intervention related to the study device including unacceptable Qp/Qs values.
Change in Qp/Qs | Baseline, 3 months, 6 months
  Comparison vs baseline of Qp/Qs value at 3 and 6 months
Change in PCWP | Baseline, 3 months, 6 months
  Comparison vs baseline of PCWP under the same test conditions